CLINICAL TRIAL: NCT03982446
Title: Prevalence of Germline Pathogenic Mutations in Patients With Pancreatic Adenocarcinoma
Brief Title: Germline Mutations in Pancreatic Adenocarcinoma
Acronym: PaMPA
Status: Completed | Type: Observational
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: Germline_pancreas
Record Dates: First submitted 2019-06-03; First posted 2019-06-11 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2020-02

CONDITIONS: Germline Mutation Abnormality; Pancreatic Cancer; Predisposition, Genetic; Hereditary Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Genetic Predisposition to Disease | interventions — Mutation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Germline DNA from white blood cells will be isolated using a commercially available blood DNA extraction kit. Remaining germline DNA will be safely stored in HeCOG's repository.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with germline mutations: This group will comprise of patients with pancreatic cancer who carry pathogenic mutations in genes associated with a predisposition to cancer.
  Interventions: Genetic: Mutations
- Patients without germline mutations: This group will comprise of patients with pancreatic cancer who did not carry pathogenic mutations in any of the genes tested, that have been previously shown to be associated with a predisposition to cancer.
  Interventions: Genetic: Mutations

INTERVENTIONS:
Genetic: Mutations

SUMMARY:
This study will assess the hereditary component of pancreatic cancer in the largest series of patients up to date through the parallel analysis of 62 cancer-associated genes. The investigators will obtain germline DNA from blood samples that have been collected from 2000 to 2019 from patients with pancreatic cancer. The investigators plan to analyze germline DNA for mutations and single nucleotide polymorphisms (SNPs) in genes that have been previously linked to a predisposition towards cancer.

The outcome can provide useful insight on the overall understanding of pancreatic pathogenesis while possible associations with age of diagnosis, tumor stage and other cancer types might arise. In addition to that, it can lead to the characterization of new variants or even new genes that predispose to pancreatic cancer.

Confirmed deleterious mutations in established cancer genes can provide valuable clinical information that can lead to effective, individualized patient management. Furthermore, family relatives of the individuals found to carry mutations can also benefit from established screening protocols for various cancer types, such as frequent colonoscopies in the case of an MMR mutation predisposing for Lynch syndrome, or preventative surgeries in the case of a deleterious BRCA1 or BRCA2 mutation. In addition to that, specific therapies that have been previously shown to be effective in breast or ovarian cancer patients with BRCA1 & BRCA2 mutations, such as platinum-based chemotherapy and PARP inhibitors can be also effective in mutations carriers with pancreatic cancer.

DETAILED DESCRIPTION:
Background Pancreatic ductal adenocarcinoma has poor prognosis mainly highlighted by the low 5-year survival rate, which is estimated to be around 6%. Although pancreatic cancer incidence is approximately 0.5% in the general population, it has a high-mortality rate. It is being registered as the fourth leading cause of cancer-related deaths in the United States. Poor prognosis is mainly attributed to the lack of efficient treatment options.

With the majority of pancreatic adenocarcinoma cases being sporadic, familial clustering (defined by the presence of at least two first degree relatives with pancreatic cancer) is observed in ~20% of the cases, whereas a clear genetic cause is identified in approximately half of these cases. Pancreatic cancer is known to occur in a range of cancer predisposing syndromes, such as hereditary breast and ovarian cancer, Peutz-Jeghers, familial adenomatous polyposis, Lynch, Li-Fraumeni and familial atypical multiple mole syndromes, while there have been clear associations with loss-of-function mutations in non-syndromic cancer genes, such as PALB2 and ATM. In addition, individuals carrying mutations in PRSS1 gene that predisposes for hereditary pancreatitis are also considered to be at high-risk for pancreatic cancer. It is therefore clear that pancreatic cancer is not related with a single cancer predisposition gene, but with numerous known and probably yet to be discovered, cancer susceptibility genes.

On the other hand, the accurate fraction of genetic predisposition in pancreatic cancer hasn't been determined. Previous studies have evaluated the prevalence of loss-of-function mutations in known cancer predisposition genes in pancreatic cancer patients through the use of multi-gene panels. The mutation yield ranged from 3.8% to 9.7% in genes that were previously found relevant to pancreatic cancer predisposition.

Through these studies, it has been highlighted that family history and stage of pancreatic cancer or age at diagnosis is not always a predictor of an underlying genetic factor, while phenotypic heterogeneity is usually associated with mutation status. The search for novel predisposition genes in pancreatic cancer patients without family history is ongoing through candidate genes analysis or through whole exome sequencing.

Research methodology Clinicopathological characteristics

Genomic DNA from pancreatic cancer patients will be retrospectively and prospectively collected from the Hellenic Cooperative Oncology Group (HeCOG) Tumor Repository, through years 2000-2019. Written informed consent has already been obtained from all patients for the use and storage of their biologic material along with their approval for their participation in research studies. The study will be in agreement with the 1975 Helsinki statement, revised in 1983.

Clinicopathologic characteristics of patients with pancreatic cancer will be retrieved form their medical record. Diagnosis will be confirmed through pathology reports, which will also provide information about grade, proliferation rate, histological subtype and lymphovascular invasion. From the patient medical record, tumor size, nodal involvement as well as metastatic lesions (TNM staging) will be reported. Importantly, detailed family history will be collected. The collection of these information will be in compliance with the regulations of the Bioethics committees of participating hospitals. Clinicopathological characteristics will be correlated with the different genomic abnormalities identified by sequencing.

Germline DNA extraction

Blood samples will be collected from patients with pancreatic cancer. Germline DNA from white blood cells will be isolated using a commercially available blood DNA extraction kit. Germline DNA will then be subjected to mechanical fragmentation via sonication to reach a DNA size of approximately 200-250 bp for downstream next-generation sequencing (NGS) analysis.

Next-Generation Sequencing

Targeted capture enrichment NGS relies on in-solution hybridization of DNA libraries with TACS (Targeted Capture Enrichment Sequences) for the identification of germline mutations in cancer patients. First, TACS that target mutations associated with hereditary cancer (in a total of 62 cancer predisposing genes) are designed and prepared by PCR followed by biotinylation. Biotinylated TACS will then be immobilized on streptavidin coated magnetic beads for subsequent hybridisation with the DNA libraries. DNA libraries are prepared from patient derived-germline DNA that fulfill quality control criteria (DNA yield, DNA integrity and fragment size) according to established protocols. Library preparation involves the 3' end and 5' end adaptor ligation and each DNA library will be barcoded using unique oligonucleotide DNA sequences to allow subsequent discrimination after sequencing. Subsequent to barcoding, samples will undergo hybridization using custom made 5'-biotynylated TACS followed by PCR amplification. Finally, enriched DNA libraries will be normalised and pooled on a NGS platform prior to paired-end sequencing using manufacturer's protocols.

Bioinformatic and Data Analysis Sequence data from leucocyte (buffy coat) DNA will be demultiplexed and aligned to the human genome (hg19) using appropriate aligner algorithms (BWA) to generate a BAM file. A combination of variant calling algorithms will be used to call germline mutations. Local realignment will be performed for accurate detection of small insertions and deletions and appropriate algorithms to detect rearrangements. Bioinformatics tools for copy number alterations (CNAs) calling such as ASCAT-2, CNVkit or ANACONDA will be used for the assessment of focal gene amplification or deletion events. Read depth-based analysis will also be taken into consideration for assessment of gene-level CNAs. Appropriate variant annotators will be used to annotate the identified alterations to each gene. Germline variant databases such as ClinVar will be used for the classification of variants according to the ACMG guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with adenocarcinoma of the pancreas
* All disease stages

Exclusion criteria

* Patients with pancreatic cancer, other than adenocarcinoma
* Non-eligible blood samples

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Genomic DNA from patients with pancreatic cancer will be retrospectively and prospectively collected from the Hellenic Cooperative Oncology Group (HeCOG) Tumor Repository, through years 2000-2019. Written informed consent has already been obtained from all patients for the use and storage of their biologic material along with their approval for their participation in research studies. The study will be in agreement with the 1975 Helsinki statement, revised in 1983.
Sampling Method: Non-Probability Sample
Enrollment: 549 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Time Frame: through the completion of the study, up to 2 years
  Evaluation of overall survival in patients with pancreatic cancer, from the date of treatment start until verified disease progression, death from any cause or date of last contact whichever occurred first

CONTACTS AND LOCATIONS:
Locations (1):
- Hellenic Oncology Cooperative Group, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fountzilas E, Eliades A, Koliou GA, Achilleos A, Loizides C, Tsangaras K, Pectasides D, Sgouros J, Papakostas P, Rallis G, Psyrri A, Papadimitriou C, Oikonomopoulos G, Ferentinos K, Koumarianou A, Zarkavelis G, Dervenis C, Aravantinos G, Bafaloukos D, Kosmidis P, Papaxoinis G, Theochari M, Varthalitis I, Kentepozidis N, Rigakos G, Saridaki Z, Nikolaidi A, Christopoulou A, Fostira F, Samantas E, Kypri E, Ioannides M, Koumbaris G, Fountzilas G, Patsalis PC. Clinical Significance of Germline Cancer Predisposing Variants in Unselected Patients with Pancreatic Adenocarcinoma. Cancers (Basel). 2021 Jan 8;13(2):198. doi: 10.3390/cancers13020198. PMID 33429865